CLINICAL TRIAL: NCT04788524
Title: Neural Correlates of Stress and Perceived Control in Adolescent Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Emily L. Belleau, Principal Investigator, Mclean Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: K23MH122668 (NIH)
Record Dates: First submitted 2021-03-03; First posted 2021-03-09 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Major Depressive Disorder
Keywords: stress; perceived control; neuroimaging; depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Intervention Model Description: Case-Control Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Computer Task Manipulation (Experimental): Participants will complete computer tasks while undergoing an fMRI brain scan
  Interventions: Behavioral: Computer Task Manipulation

INTERVENTIONS:
Behavioral: Computer Task Manipulation — Participants will complete computer tasks.

SUMMARY:
Lack of perceived control, particularly during stress, has been critically implicated in major depressive disorder (MDD) and anhedonic symptoms, especially among female adolescents; yet the neural underpinnings of perceived control disruptions in MDD remain poorly understood. Using functional magnetic resonance imaging with a novel "value of control task" in conjunction with a prospective design, this study will provide a comprehensive understanding of stress and perceived control related mechanisms in female adolescents with MDD and will examine stress-induced disruptions in perceived control as a predictor of "real world" expressions of maladaptive coping and anhedonia.

DETAILED DESCRIPTION:
Participants in this research will include 40 female adolescents, aged 14-18, with Major Depressive Disorder (MDD) and 40 healthy adolescents from the greater Boston area by Dr. Emily Belleau, at McLean Hospital's Center for Depression, Anxiety and Stress Research.

The study will include four sessions:

* A clinical diagnostic interview as well as filling out a series of questionnaires and assessments.
* The second session will include a functional magnetic resonance imaging (fMRI) brain scan to be conducted at the McLean Hospital Imaging Center. Participants will be asked to respond to surveys on their cell phone in the week following the fMRI brain scan.
* The third session will include a diagnostic interview, assessments, and questionnaires to be completed three-months after the fMRI brain scan. Participants will be asked to complete surveys on their cell phone during the week following this three month follow-up session.
* The fourth session will include a diagnostic interview, assessments, and questionnaires to be completed six-months after the fMRI brain scan. Participants will be asked to complete surveys on their cell phone during the week following this six month follow-up session.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria: All Participants

  1. Females of all ethnic origins See Section: Inclusion of Women and Minorities);
  2. Ages 14-18 (See Section: Inclusion of Children);
  3. Written informed assent/consent from adolescent and parent/guardian (if under age 18);
  4. English as a first language or English fluency;
  5. Right handed111;
  6. Personal cell-phone (for Ecological Momentary Assessment [EMA]) 7 All participants will be in the follicular phase of their menstrual cycle when completing the functional magnetic resonance imaging (fMRI) study session

Inclusion Criteria: MDD Sample

1. Meet Diagnostic Statistical Manual-5th edition (DSM-5) diagnostic criteria for major depressive disorder (as diagnosed with the KSADS)
2. Absence of any psychotropic medications for at least 2 weeks (6 weeks for fluoxetine; 6 months for neuroleptics; 2 weeks for benzodiazepines; 2 weeks for any other antidepressants);

Inclusion Criteria: Healthy Control (HC) Sample

1. No history or current diagnosis of any DSM-5 psychiatric or substance/alcohol-related disorder (as diagnosed with the KSADS)
2. No first-degree relatives with a history of depression, bipolar disorder, or psychosis

Exclusion Criteria:

* Exclusion Criteria: All Participants

  1. History of head trauma with loss of consciousness;
  2. History of seizure disorder;
  3. Serious or unstable medical illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurologic or hematologic disease;
  4. History of cocaine or stimulant use (e.g., amphetamine, cocaine, methamphetamine);
  5. History of use of dopaminergic drugs (including methylphenidate);
  6. Use of hormonal replacement therapy, anabolic steroids, or hormonal contraception;
  7. Clinical or laboratory evidence of hypothyroidism;
  8. Systemic medical or neurological illness that could impact fMRI measures of cerebral blood flow;
  9. Failure to meet standard exclusion criteria for fMRI scanning (e.g., claustrophobia, cardiac pacemakers, neural pacemakers, surgically implanted metal devices, cochlear implants, metal braces, or other metal objects in the body);
  10. Pregnancy
  11. Testing positive on a drug test on the day of the scan which testis for stimulants, marijuana, barbiturates, benzodiazepine, buprenorphine, 3,4-Methyl enedioxy methamphetamine (MDMA), methadone, opiates, oxycodone, phencyclidine;
  12. History of electroconvulsive therapy
  13. Participants with suicidal ideation where study participation is deemed unsafe by the study clinician;

Additional Exclusion Criteria: Major Depressive Disorder (MDD) Sample

1. Major depressive disorder diagnosis secondary to another disorder (selected comorbid anxiety disorders such as generalized anxiety disorder, specific phobia, and social anxiety disorders are allowed if they are secondary to MDD)

Ages: 14 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Only female.
Enrollment: 80 (Estimated)
Dates: Start 2021-04-23 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Blood-Oxygen-Level-Dependent Imaging (BOLD) activation of the ventral striatum and ventral medial prefrontal cortex | 1.5 hour long scan during session 2
  BOLD activation of frontostriatal regions in response to computer tasks performed during the fMRI Brian scan

SECONDARY OUTCOMES:
Cortisol Rating | collected as part of 1.5 hour long scan during session 2
  Saliva rating to be collected throughout the fMRI brain scan
Mood Rating | collected as part of 1.5 hour long scan during session 2
  Self-reported mood rating to be collected throughout the fMRI brain scan
Stress Reactivity Score | Longitudinal, three time points (baseline, 3-month follow-up, 6-month follow-up)
  Stress Reactivity Survey Item collected via smart-phone delivered ecological momentary assessment
Stress Reactive Rumination Score | Longitudinal, three time points (baseline, 3-month follow-up, 6-month follow-up)
  Stress Reactive Rumination Scale collected via smart-phone delivered ecological momentary assessment
Positive Affect Score | Longitudinal, three time points (baseline, 3-month follow-up, 6-month follow-up)
  Positive Affect Survey Items collected via smart-phone delivered ecological momentary assessment

CONTACTS AND LOCATIONS:
Overall Officials: Emily L Belleau, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No